CLINICAL TRIAL: NCT05098041
Title: A Phase 1 Open-Label Study to Evaluate the Drug-Drug Interaction of Rifampin as a Strong CYP3A Inducer on Soticlestat Pharmacokinetics in Healthy Adult Participants
Brief Title: A Study of Soticlestat and Rifampin in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: TAK-935-1009
Record Dates: First submitted 2021-10-20; First posted 2021-10-28 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — soticlestat; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Soticlestat 300 mg + Rifampin 600 mg (Experimental): Soticlestat 3*100 mg tablets, orally, administered once on Day 1 in fasted state in Period 1, followed by a washout period of 4 days, further followed by Rifampin 600 mg, administered as 2*300mg capsules, orally, once daily for 13 consecutive days, from Day 1 to Day 13 in fasted state in Period 2. Soticlestat 3*100 mg tablets, will be administered orally along with rifampin 600 mg (2*300mg) capsules, orally in the morning of Day 11 in Period 2.
  Interventions: Drug: Soticlestat; Drug: Rifampin

INTERVENTIONS:
Drug: Soticlestat — Soticlestat tablets.
  Other Names: TAK-935
Drug: Rifampin — Rifampin capsules.

SUMMARY:
The main aim of this study is to check how rifampin affects the way soticlestat is processed by the body.

Participants will be required to stay at the study clinic for 18 consecutive days. On the first full day and 15th day, participants will take a single dose of soticlestat. Rifampin will be taken each day starting on the 5th day for 13 consecutive days.

Clinic staff will follow up with each participant about 15 days after the last soticlestat dose to check for any side effects.

DETAILED DESCRIPTION:
The drug being tested in this study is called soticlestat (TAK-935). The study will evaluate the safety and tolerability of soticlestat when co-administered with rifampin in healthy participants.

The study will enroll 14 participants. The participants will be assigned to treatment group to receive following therapies:

• Soticlestat 300 milligram (mg) + Rifampin 600 mg

The study will have two periods: Period 1 and Period 2. In Period 1, participants will receive soticlestat in fasted condition while in Period 2 participants will receive soticlestat along with rifampin. The data will be collected and stored in electronic case report form (eCRF).

This single-center trial will be conducted in the United Kingdom. The overall study duration of the study will be approximately 58 days including 28 days screening and follow up duration. There will be a follow up contact required for all participants approximately 15 days after the last dose of soticlestat.

ELIGIBILITY:
Inclusion criteria:

1. Healthy, adult, male or female of non-childbearing potential, 18-55 years of age, inclusive, at screening.
2. Has body mass index (BMI) greater than or equal to (>=) 18.0 and less than or equal to (<=) 32.0 kilogram per square meter (kg/m^2) at screening.
3. Continuous non-smoker who has not used nicotine-containing products for at least 90 days prior to the first dosing.
4. Able to swallow multiple tablets/capsules.

Exclusion criteria:

1. Has history of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
2. Any positive responses on the C-SSRS that in the clinical judgment of the Investigator has a risk of suicide or has made a suicide attempt in the previous 12 months prior to the first dosing.
3. Unable to refrain from or anticipates the use of:

   * Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing. Thyroid hormone replacement medication may be permitted if the participant has been on the same stable dose for the immediate 3 months prior to first dosing.
   * Any drugs known to be significant inducers of cytochrome (CYP)3A, CYP2C19, UGT1A9 or UGT2B4 enzymes, and/or P-glycoprotein (P-gp), including St. John's Wort, within 28 days prior to the first dosing.

   Appropriate sources (example, Flockhart TableTM) will be consulted to confirm lack of pharmacokinetic (PK)/pharmacodynamics interaction with study drug.
4. History of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to the following: beer 354 milliliter [mL]/12 ounce [oz], wine [118 mL/4 oz], or distilled spirits [29.5 mL/1 oz] per day).
5. Consumes excessive amounts, defined as greater than 4 servings (1 serving is approximately equivalent to 120 mg of caffeine), of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
6. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
7. Donation of blood or significant blood loss within 56 days prior to the first dosing.
8. Plasma donation within 7 days prior to the first dosing.
9. Participation in another clinical study within 30 days or 5 half-lives prior to the first dosing. The 30-days window or 5 half-lives will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/6181d800eb0e19002afd69ec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in United Kingdom from 22 November 2021 to 03 March 2022.
Pre-assignment Details: Healthy participants were enrolled in this 2-period study to receive soticlestat tablets alone in Period 1 and soticlestat tablets and rifampin capsules in Period 2 of the study.
Groups:
- All Participants: Soticlestat 300 mg + Rifampin 600 mg + Soticlestat 300 mg: Soticlestat 300 milligram (mg) (3*100 mg) immediate-release (T4) tablet, orally, once on Day 1 in fasted state in Period 1, followed by a washout period of 4 days, further followed by Rifampin 600 mg (2*300 mg), capsules, orally, once daily from Day 1 to Day 13 along with soticlestat 300 mg (3*100 mg) T4 tablet, orally, once on Day 11 in fasted state in Period 2.
Period: Period 1 (1 Day)
Arm/Group | All Participants: Soticlestat 300 mg + Rifampin 600 mg + Soticlestat 300 mg
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Washout Period (4 Days)
Arm/Group | All Participants: Soticlestat 300 mg + Rifampin 600 mg + Soticlestat 300 mg
Started | 14
Completed | 14
Not Completed | 0
Period: Period 2 (13 Days)
Arm/Group | All Participants: Soticlestat 300 mg + Rifampin 600 mg + Soticlestat 300 mg
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received at least one dose of the study drug(s).
Groups:
- All Participants: Soticlestat 300 mg + Rifampin 600 mg + Soticlestat 300 mg: Soticlestat 300 mg (3*100 mg) immediate-release (T4) tablet, orally, once on Day 1 in fasted state in Period 1, followed by a washout period of 4 days, further followed by Rifampin 600 mg (2*300 mg), capsules, orally, once daily from Day 1 to Day 13 along with soticlestat 300 mg (3*100 mg) T4 tablet, orally, once on Day 11 in fasted state in Period 2.
Arm/Group | All Participants: Soticlestat 300 mg + Rifampin 600 mg + Soticlestat 300 mg
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (10.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 15
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 173.9 (5.73)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 80.72 (10.176)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 26.713 (3.1941)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Soticlestat When Administered Alone and With Rifampin
Time Frame: Soticlestat Alone: Day 1 pre-dose and at multiple timepoints (up to 96 hours) post-dose in Period 1; Soticlestat with Rifampin: Day 11 pre-dose and at multiple time points (up to 72 hours) post-dose in Period 2
Population: The pharmacokinetic (PK) set included participants who complied sufficiently with the protocol and display an evaluable PK profile (example, exposure to treatment, availability of measurements and absence of major protocol violations).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Soticlestat 300 mg Alone: Soticlestat 300 mg (3*100 mg) T4 tablet, orally, once on Day 1 in fasted state in Period 1.
- Soticlestat 300 mg + Rifampin 600 mg: Rifampin 600 mg (2*300 mg), capsules, orally, once daily from Day 1 to Day 13 along with soticlestat 300 mg (3*100 mg) T4 tablet, orally, once on Day 11 in fasted state in Period 2.
Arm/Group | Soticlestat 300 mg Alone | Soticlestat 300 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
nanogram per milliliter (ng/mL) | 1364 (63.6) | 176.8 (99.6)
Statistical Analysis 1: Comparison: Soticlestat 300 mg Alone vs Soticlestat 300 mg + Rifampin 600 mg; Test type: Other — Linear mixed-effects model was used for analysis. The model included treatment as a fixed effect and participant as a random effect. The point estimates and 90 percent (%) confidence intervals (CIs) for the Geometric Mean Ratio (GMR) of Cmax for Soticlestat and Rifampin versus Soticlestat alone were calculated using the exponentiation of the point estimates of the difference between treatment regimen and the corresponding 90% CIs from the analyses on the natural-log (ln)-transformed Cmax; Geometric Mean Ratio (%) = 13.15, 90% CI 2-sided [9.73 to 17.79] — GMR (%) was calculated as 100*(Soticlestat + Rifampin/Soticlestat Alone)

2. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Soticlestat When Administered Alone and With Rifampin
Time Frame: as for outcome 1
Population: The PK set included participants who complied sufficiently with the protocol and display an evaluable PK profile (example, exposure to treatment, availability of measurements and absence of major protocol violations). Here, "overall number of participants analyzed" signified those who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter(ng*hr/mL)
Groups:
- Soticlestat 300 mg Alone: Soticlestat 300 mg administered as 3*100 mg tablets, orally, administered once on Day 1 in fasted state in Period 1.
Arm/Group | Soticlestat 300 mg Alone | Soticlestat 300 mg + Rifampin 600 mg
Number analyzed (Participants) | 13 | 11
nanogram*hour per milliliter(ng*hr/mL) | 1448 (47.0) | 226.2 (94.0)
Statistical Analysis 1: Comparison: Soticlestat 300 mg Alone vs Soticlestat 300 mg + Rifampin 600 mg; Test type: Other — Linear mixed-effects model was used for analysis. The model included treatment as a fixed effect and participant as a random effect. The point estimates and 90% CIs for the GMR of AUC∞ for Soticlestat and Rifampin versus Soticlestat alone were calculated using the exponentiation of the point estimates of the difference between treatment regimen and the corresponding 90% CIs from the analyses on the ln-transformed AUC∞; Geometric Mean Ratio (%) = 16.42, 90% CI 2-sided [12.53 to 21.50] — GMR (%) was calculated as 100*(Soticlestat + Rifampin/Soticlestat Alone)

3. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Soticlestat When Administered Alone and With Rifampin
Time Frame: as for outcome 1
Population: The PK set included participants who complied sufficiently with the protocol and display an evaluable PK profile (example, exposure to treatment, availability of measurements and absence of major protocol violations).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Soticlestat 300 mg Alone | Soticlestat 300 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
ng*hr/mL | 1290 (52.9) | 190.6 (88.2)
Statistical Analysis 1: Comparison: Soticlestat 300 mg Alone vs Soticlestat 300 mg + Rifampin 600 mg; Test type: Other — Linear mixed-effects model was used for analysis. The model included treatment as a fixed effect and participant as a random effect. The point estimates and 90% CIs for the GMR of AUClast for Soticlestat and Rifampin versus Soticlestat alone were calculated using the exponentiation of the point estimates of the difference between treatment regimen and the corresponding 90% CIs from the analyses on the ln-transformed AUClast; Geometric Mean Ratio (%) = 14.92, 90% CI 2-sided [11.94 to 18.64] — GMR (%) was calculated as 100*(Soticlestat + Rifampin/Soticlestat Alone)

4. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Soticlestat When Administered Alone and With Rifampin
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Soticlestat 300 mg Alone | Soticlestat 300 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
hour | 0.504 [0.24 to 0.76] | 0.499 [0.27 to 0.75]
Statistical Analysis 1: Comparison: Soticlestat 300 mg Alone vs Soticlestat 300 mg + Rifampin 600 mg; Test type: Other; p = 0.07910, Wilcoxon Signed-Rank Test; Median Difference (Final Values) = -0.117, 90% CI 2-sided [-0.202 to 0.000] — Difference was calculated as (Soticlestat + Rifampin) - Soticlestat Alone. The difference of medians (treatment effect) and the corresponding 90% CI was estimated using the Hodges-Lehmann method and Walsh Averages

5. Secondary Outcome: Number of Participants Reported One or More Treatment-Emergent Adverse Events (TEAEs)
Time Frame: From Day 1 of Period 1 up to 15 days after the last dose of Soticlestat in Period 2 (up to Day 31)
Population: The safety set included all participants who received at least one dose of the study drug(s).
Measure: Count of Participants; unit: Participants
Groups:
- Rifampin 600 mg Alone: Rifampin 600 mg (2*300 mg), capsules, orally, once daily from Day 1 to Day 13 in fasted state in Period 2.
Arm/Group | Soticlestat 300 mg Alone | Rifampin 600 mg Alone | Soticlestat 300 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14 | 14
Participants | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: TEAEs were adverse events (AE) that started from Day 1 of Period 1 up to 15 days after the last dose of Soticlestat in Period 2 (up to Day 31)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Soticlestat 300 mg Alone | Rifampin 600 mg Alone | Soticlestat 300 mg + Rifampin 600 mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 2/15 | 1/14 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Soticlestat 300 mg Alone (N=15) | Rifampin 600 mg Alone (N=14) | Soticlestat 300 mg + Rifampin 600 mg (N=14)
Bacteriuria (Infections and infestations) | 1 | 0 | 0
Catheter site erythema (General disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT05098041/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT05098041/SAP_001.pdf